CLINICAL TRIAL: NCT01043523
Title: An Observational Study of the Administration of Eovist/Primovist in Pediatric Subjects (> 2 Months and Less Than 18 Years) Who Are Referred for a Routine Contrast Enhanced Liver MRI Because of Suspected or Known Focal Liver Lesions
Brief Title: Liver MRI With Primovist/Eovist in Pediatric Subjects Who Are Suspected or Have Focal Liver Lesions.
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 13729
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Liver Neoplasms; Adenoma; Carcinoma; Liver Abscess
Keywords: Liver neoplasms; Adenoma; Liver cell carcinoma; Hepatocellular; Liver abscess
MeSH Terms: conditions — Liver Neoplasms; Adenoma; Carcinoma; Liver Abscess; Carcinoma, Hepatocellular | interventions — gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Pediatric subjects who have had a Eovist/Primovist enhanced MRI for known or suspected focal liver disease
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Gadoxetic Acid Disodium (Eovist, BAY86-4873)

INTERVENTIONS:
Drug: Gadoxetic Acid Disodium (Eovist, BAY86-4873) — Participants have received Primovist/Eovist for liver Magnetic Resonance Imaging (MRI) as part of their routine care at participating institutions and additional diagnostic information are identified retrospectively from institution records

SUMMARY:
Medical records are reviewed to obtain information about the use of a MRI diagnostic imaging agent (contrast agent) called Primovist/Eovist in children older than 2 months and less than 18 years. Data that has been recorded in the child's medical records relating to the injection of Primovist/Eovist will be collected. Information will be collected from up to 2 weeks before the child received Primovist/Eovist until 12 months after the child received Primovist/Eovist. Copy of the child's MR images that were taken right before and after the child received Primovist/Eovist and all other reports (laboratory reports, other imaging reports, etc) that are part of the child's medical records during that time period will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age >2 months and <18 years of age at the time of the Primovist/Eovist enhanced MRI
* MRI with Primovist/Eovist due to suspected or known focal liver lesions
* Evaluable safety data
* Evaluable efficacy data: precontrast and postcontrast magnetic resonance (MR) images must be available for review
* If the above criteria are met, the principal investigator (PI) and/or designee will obtain a signed consent for medical records release including access to anonymized electronic copies of the pre- and post-Primovist/Eovist MRI scans, in accordance with local regulatory requirements in order for subjects to be enrolled in the study.

Exclusion Criteria:

* A subject will be excluded from this observational / retrospective study if the subject has previously been enrolled into this study. Subjects may only be entered once into this study, even if they have been imaged multiple times and for different indications.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric subjects who have had a Primovist/Eovist enhanced MRI for known or suspected focal liver disease
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2009-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- United States (5):
  - Palo Alto, California
  - New York, New York
  - Durham, North Carolina
  - Cinncinati, Ohio
  - Hershey, Pennsylvania
- Many Locations, Italy
- Many Locations, Japan
- Many Locations, Singapore
- Many Locations, Taiwan

REFERENCES:
- [Result] Geller J, Kasahara M, Martinez M, Soresina A, Kashanian F, Endrikat J. Safety and Efficacy of Gadoxetate Disodium-Enhanced Liver MRI in Pediatric Patients Aged >2 Months to <18 Years-Results of a Retrospective, Multicenter Study. Magn Reson Insights. 2016 Jul 21;9:21-8. doi: 10.4137/MRI.S39091. eCollection 2016. PMID 27478381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric subjects (> 2 months and < 18 years of age), who underwent a contrast-enhanced (CE) liver magnetic resonance imaging (MRI) with Eovist/Primovist because of suspected or known focal liver lesions, and who had evaluable safety and efficacy data.
Pre-assignment Details: Of the 52 subjects that were identified by the investigators for participation in this observational/retrospective study, 51 were included in the efficacy analysis. One subject (22001-0005) did not have unenhanced images. The safety analysis was performed on all 52 subjects.
Period: Overall Study
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Started | 52
Participants With Unenhanced Images | 51
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 52
Age, Customized [Number; unit: Participants]
  >2 months to ≤2 years | 14
  >2 years to ≤12 years | 25
  >12 years to <18 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 24
Indication for magnetic resonance imaging (MRI) [Number; unit: Participants]
  Suspected or known focal liver lesions | 49
  Cystic fibrosis | 1
  Biliary atresia | 1
  No clinical indication | 1
Physical examination performed at preinjection timepoint [Number; unit: Participants] — Number of participants received physical examination within14 days prior to injection.
  Participants
    Yes | 36
    No | 16
Physical examination performed at postinjection timepoint [Number; unit: Participants] — Number of participants received physical examination up to 24 hours after injection of Eovist/Primovist. Changes in the physical examination were recorded as adverse events (AEs).
  Participants
    Yes | 35
    No | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Change in Additional Diagnostic Information Obtained When Comparing the Combined Precontrast/Postcontrast Images With the Precontrast Images.
Description: Overall Change in additional diagnostic information was defined as a change in at least 1 of the 5 variables below obtained from the combined precontrast and postcontrast images as compared with the precontrast images: 1. Change in number of lesions: greater or fewer 2. Improved border delineation of the primary lesion 3. Increased contrast of primary lesion versus. background 4. Change in size of the primary lesion: larger or smaller 5. Change in information about lesion characterization (lesion type): improved, unchanged, worsened
Time Frame: When precontrast and postcontrast images are available from all enrolled subjects, on average 1 year post Primovist/Eovist MRI
Population: Analysis is based on subjects with available precontrast and combined precontrast/postcontrast images (n=51)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 51
Percentage of participants | 86.3 [73.7 to 94.3]

2. Primary Outcome: Number of Participants With Laboratory Values Considered to be Clinically Relevant Values or Abnormalities at Pre-injection Time Point
Description: Laboratory parameters analyzed: Hematology: leukocytes, erythrocytes, hematocrit, platelets, hemoglobin, prothrombin time and differential counts (neutrophils total, neutrophils segmented and lymphocytes); Chemistry: lactate dehydrogenase (LDH), alkaline phosphatase (AKP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), sodium, potassium, blood urea nitrogen (BUN), glucose, creatinine, bilirubin:, direct bilirubin, indirect bilirubin, total protein, albumin, estimated glomerular filtration rate (eGFR), and α-fetoprotein levels.
Time Frame: 14 days prior to Eovist/Primovist MRI
Population: The laboratory analyses were performed on participants in the Full Analysis Set (FAS) who had laboratory values collected
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 40
Participants
  Increased AST, BUN | 1
  Increased AST, AKP | 1
  High liver values due to gastrointestinal (GI) | 1

3. Primary Outcome: Number of Participants With Laboratory Values Considered to be Clinically Relevant Values or Abnormalities 24 Hours Post-injection
Description: The following parameters were analyzed: Hematology: leukocytes, erythrocytes, hematocrit, platelets, hemoglobin, prothrombin time and differential counts (neutrophils total, neutrophils segmented and lymphocytes) Clinical chemistry: lactate dehydrogenase (LDH), alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), sodium, potassium, blood urea nitrogen (BUN), glucose, creatinine, total bilirubin, direct bilirubin, indirect bilirubin, total protein, albumin, eGFR, and α-fetoprotein levels.
Time Frame: Up to 24 hours post-Eovist/Primovist MRI
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 30
Participants | 0

4. Primary Outcome: Vital Signs: Mean Change From Baseline in Heart Rate
Time Frame: 14 days prior to and up to 24 hours post-Eovist/Primovist MRI
Population: The vital signs analyses were performed on participants in the Full Analysis Set (FAS) who had vital signs collected both precontrast and postcontrast
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 30
beats/min | -4.17 (16.86)

5. Primary Outcome: Vital Signs: Mean Change From Baseline in Systolic Blood Pressure
Time Frame: 14 days prior to and up to 24 hours post-Eovist/Primovist MRI
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 25
mmHg | -1.76 (17.10)

6. Primary Outcome: Vital Signs: Mean Change From Baseline in Diastolic Blood Pressure
Time Frame: 14 days prior to and up to 24 hours post-Eovist/Primovist MRI
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 24
mmHg | -0.46 (17.00)

7. Secondary Outcome: Change in Diagnosis Obtained From the Combined Precontrast and Postcontrast Images as Compared With the Precontrast Images
Time Frame: as for outcome 1
Population: Analysis is based on subjects with available precontrast and combined precontrast/postcontrast images (n=51)
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 51
Participants
  Relevant change in diagnosis | 25
  No change in diagnosis | 26

8. Secondary Outcome: Change in Confidence of Diagnosis Obtained From the Combined Precontrast and Postcontrast Images as Compared With the Precontrast Images
Time Frame: as for outcome 1
Population: Analysis is based on subjects with available precontrast and combined precontrast/postcontrast images (n=51)
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 51
Participants
  Blinded reader was confident in the diagnosis | 10
  Blinded reader was not confident in the diagnosis | 41

9. Secondary Outcome: Change in Number of Nonmalignant Lesions Obtained From the Combined Precontrast and Postcontrast Images as Compared With the Precontrast Images
Description: Change in number of nonmalignant lesions was defined as a change from more to less or less to more obtained from the combined precontrast and postcontrast images as compared with the precontrast images
Time Frame: as for outcome 1
Population: Analysis is based on subjects with available precontrast and combined precontrast/postcontrast images (n=51)
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 51
Participants
  Change in the number of non-malignant lesions | 18
  No change in the number of non-malignant lesions | 33

10. Secondary Outcome: Change in Number of Malignant Lesions Obtained From the Combined Precontrast and Postcontrast Images as Compared With the Precontrast Images
Description: Change in number of malignant lesions was defined as a change from more to less or less to more obtained from the combined precontrast and postcontrast images as compared with the precontrast images
Time Frame: as for outcome 1
Population: Analysis is based on subjects with available precontrast and combined precontrast/postcontrast images (n=51)
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 51
Participants
  Change in the number of malignant lesions | 11
  No change in the number of malignant lesions | 40

11. Secondary Outcome: Change in Recommended Next Course of Subject Management/Therapy Obtained From the Combined Precontrast and Postcontrast Images as Compared With the Precontrast Images
Time Frame: as for outcome 1
Population: Analysis is based on subjects with available precontrast and combined precontrast/postcontrast images (n=51)
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 51
Participants
  Change from subject management therapy | 45
  No change in subject management therapy | 6

12. Secondary Outcome: Change in Recommended Next Course of Subject Management / Therapy - Comparison of Precontrast Versus Combined Precontrast/Postcontrast Images (Only Subjects for Whom a Change Was Documented)
Time Frame: as for outcome 1
Population: 45 subjects had a change from additional imaging with contrast-enhanced MRI based on the precontrast images to definitive therapy.
Measure: Number; unit: Participants
Groups:
- Precontrast: 45 subjects had a change based on the Precontrast image read
- Combined Precontrast / Postcontrast: Based on the Combined precontrast / postcontrast image read, biopsy was recommended for 24 subjects and follow-up for 13 subjects
Arm/Group | Precontrast | Combined Precontrast / Postcontrast
Number analyzed (Participants) | 45 | 45
Participants
  Ultrasound | 7 | 1
  Biopsy | 0 | 26
  Follow-up examination | 1 | 13
  Other | 37 | 2
  No action | 0 | 3

13. Secondary Outcome: The Overall Image Quality for the Postcontrast Image Only
Time Frame: as for outcome 1
Population: Analysis is based on subjects with available precontrast and combined precontrast/postcontrast images (n=51)
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 51
Participants
  Satisfactory | 34
  Excellent | 8
  Poor | 9

14. Secondary Outcome: Final Diagnosis (SoT) by Clinical Investigator
Time Frame: as for outcome 1
Population: Analysis is based on subjects with available precontrast and combined precontrast/postcontrast images (n=51)
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 51
Participants
  Benign Lesions | 27
  Malignant Lesions | 24

15. Secondary Outcome: Sensitivity, Specificity and Accuracy of Blinded Read of Precontrast and Combined Precontrast/Postcontrast Images Based on Final Diagnosis.
Description: Sensitivity is the probability that a test indicates there is disease when there is disease. Specificity is the probability that a test indicates there is no disease when there is no disease. Accuracy is the probability that a test is correct: the test indicates there is no disease when there is no disease and it indicates there is disease when there is disease.
Time Frame: as for outcome 1
Population: Analysis is based on subjects with available precontrast and combined precontrast/postcontrast images (n=51)
Measure: Number; unit: Percentage points
Groups:
- Precontrast; Combined Precontrast / Postcontrast: 51 eligible for accuracy, 24 eligible for sensitivity, 27 eligible for specificity
Arm/Group | Precontrast | Combined Precontrast / Postcontrast
Number analyzed (Participants) | 51 | 51
Percentage points
  Sensitivity [%] | 66.7 | 70.8
  Specificity [%] | 88.9 | 66.7
  Accuracy [%] | 78.4 | 68.6

16. Other Pre Specified Outcome: Change in Number of Lesions Obtained From the Combined Precontrast and Postcontrast Images as Compared With the Precontrast Images
Time Frame: as for outcome 1
Population: Analysis is based on subjects with available precontrast and combined precontrast/postcontrast images (n=51)
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 51
Participants
  Less | 3
  Equal | 34
  More | 14

17. Other Pre Specified Outcome: Improved Border Delineation of the Primary Lesion Obtained From the Combined Precontrast and Postcontrast Images as Compared With the Precontrast Images
Time Frame: as for outcome 1
Population: Analysis is based on subjects with available precontrast and combined precontrast/postcontrast images (n=51)
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 51
Participants
  Yes | 36
  No | 15

18. Other Pre Specified Outcome: Increased Contrast of Primary Lesion vs Background Obtained From the Combined Precontrast and Postcontrast Images as Compared With the Precontrast Images
Time Frame: as for outcome 1
Population: Analysis is based on subjects with available precontrast and combined precontrast/postcontrast images (n=51)
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 51
Participants
  Yes | 40
  No | 11

19. Other Pre Specified Outcome: Change in Size of the Primary Lesion Obtained From the Combined Precontrast and Postcontrast Images as Compared With the Precontrast Images
Time Frame: as for outcome 1
Population: Analysis is based on subjects with available precontrast and combined precontrast/postcontrast images (n=51)
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 51
Participants
  Larger | 12
  No change | 38
  Smaller | 1

20. Other Pre Specified Outcome: Change in Information About Lesion Characterization Obtained From the Combined Precontrast and Postcontrast Images as Compared With the Precontrast Images
Time Frame: as for outcome 1
Population: Analysis is based on subjects with available precontrast and combined precontrast/postcontrast images (n=51)
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Number analyzed (Participants) | 51
Participants
  Improved | 39
  Unchanged | 12
  Worsened | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 24 hours after Eovist/Primovist injection. Serious adverse event data were collected up to 1 year post the Eovist/Primovist MRI administration.
Groups:
- Gadoxetic Acid Disodium (Eovist, BAY86-4873): Participants have received Primovist/Eovist for liver MRI as part of their routine care at participating institutions and additional diagnostic information are identified retrospectively from institution records.
Arm/Group | Gadoxetic Acid Disodium (Eovist, BAY86-4873)
Serious Adverse Events (participants affected / at risk) | 21/52
Other Adverse Events (participants affected / at risk) | 1/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gadoxetic Acid Disodium (Eovist, BAY86-4873) (N=52)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Caecitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1
Gait disturbance (General disorders) | 1
Pyrexia (General disorders) | 3
Device occlusion (General disorders) | 1
Cholangitis acute (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Enterococcal bacteraemia (Infections and infestations) | 1
Gastroenteritis rotavirus (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 2
Parainfluenzae virus infection (Infections and infestations) | 1
Feeding disorder (Metabolism and nutrition disorders) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Renal tubular acidosis (Renal and urinary disorders) | 1
Portal shunt (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gadoxetic Acid Disodium (Eovist, BAY86-4873) (N=52)
Benign tumour excision (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No